CLINICAL TRIAL: NCT07238712
Title: Optimization of Post-transplantation Benadamustine and Cyclophosphamide in Patients With High-risk Myeloid Malignancies and a Partially Mismatched Donor (APTBCy)
Brief Title: Optimization of Post-transplantation Benadamustine and Cyclophosphamide in Patients With High-risk Myeloid Malignancies and a Partially Mismatched Donor
Acronym: APTBCy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, RM Gorbacheva Research Institute Scientific director, St. Petersburg State Pavlov Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30/25-n
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia (AML); Chronic Myeloid Leukemia; Myelodysplastic Syndromes (MDS); Myeloprolipherative Neoplsm; Atypical Chronic Myeloid Leukemia
Keywords: Post-transplantation cyclophosphamide; Post-transplantation bendamustine; graft-versus-host disease; abatacept; ruxolitinib
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Graft vs Host Disease | interventions — ruxolitinib; Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Test cohort 1 - ruxolitinib (Experimental): Days +3 through +4: Bendamustine 50 mg/m2 iv x 2 days; Days +3 through +4: Cyclophosphamide 25 mg/kg iv x 2 days; Days -1 through +21: ruxolitinib 10 mg/kg/day p.o.; mycophenolate mofetil Days +5 through +35 30 mg/kg/day p.o.; Days +5 through +100: Tacrolimus 0.03 mg/kg/day with further correction by concentration
  Interventions: Drug: Ruxolitinib
- Test cohort 2 - abatacept (Experimental): Days +3 through +4: Bendamustine 50 mg/m2 iv x 2 days; Days +3 through +4: Cyclophosphamide 25 mg/kg iv x 2 days; Days -1 through +21: ruxolitinib 10 mg/kg/day p.o.; mycophenolate mofetil Days +5 through +35 30 mg/kg/day p.o.; Days +5 through +100: Tacrolimus 0.03 mg/kg/day with further correction by concentration
  Interventions: Drug: Abatacept (Orencia)
- Experimental: Expansion cohort (Experimental): Days +3 through +4: Bendamustine 50 mg/m2 iv x 2 days; Days +3 through +4: Cyclophosphamide 25 mg/kg iv x 2 days; Days -1,+5, +14, +21 abatacept 10 mg/kg/day i.v.; Days +5 through +100: Tacrolimus 0.03 mg/kg/day with further correction by concentration
  Interventions: Drug: Abatacept (Orencia)

INTERVENTIONS:
Drug: Ruxolitinib — ; Days -1 through +21: ruxolitinib 10 mg/kg/day p.o.
  Arms: Experimental: Test cohort 1 - ruxolitinib
Drug: Abatacept (Orencia) — Days -1,+5, +14, +21 abatacept 10 mg/kg/day i.v.
  Arms: Experimental: Expansion cohort; Test cohort 2 - abatacept

SUMMARY:
Optimization of bendamustine-containg graft-versus-host disease (GVHD) prophylaxis to reduce the incidence of secondary haemophagocytic lymphohistiocytosis and GVHD

DETAILED DESCRIPTION:
Prognosis of patients undergoing allogeneic stem cell transplantation (HCT) for high-risk myeloid malignancies, including refractory acute myeloid leukemia, with standard HCT technologies have relatively poor prognosis with 10-30% long-term disease-free survival. One of the approaches to augment graft-versus-leukemia effect the use of post-transplantation bendamustine in graft-versus-host disease prophylaxis. Despite high frequency of responses and durable remissions after this approach majority of patients develop a serious complication - cytokine release syndrome, which can be life-threatening in some patients. The combination bendamustine (PTB) and post-transplantation cyclophosphamide (PTCY) facilitates comparable graft-versus leukemia effect to PTB, but with better safety profile and reduced incidence of severe cytokine release syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for allogeneic hematopoietic stem cell transplantation
* Patients with <10/10 HLA-matched related or unrelated donor available. The donor and recipient must be identical by the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA-DQB1.
* Peripheral blood stem cells or bone marrow as a graft source
* Diagnosis:

Acute myeloid leukemia Chronic myeloid leukemia, Ph+ Myelodysplastic Syndromes Myeloprolipherative neoplasms - High-risk disease defined as: Acute myeloid leukemia: >5% of clonal blasts in bone marrow despite adequate previous induction therapy or allogeneic stem cell transplantation Myelodysplastic Syndrome: >5% of blasts despite previous therapy Myeloid malignancy with with -7 or complex karyotype, or p53 mutation regardless of blast count in bone marrow Treatment-related myelodysplastic syndrome Second or subsequent allogeneic HCT after relapse of a myeloid malignancy Chronic myelomonocytic leukemia Myeloprolipherative neoplasms, unclassifiable

- No severe concurrent illness

Exclusion Criteria:

* Patients with indication for allogeneic hematopoietic stem cell transplantation
* Patients with <10/10 HLA-matched related or unrelated donor available. The donor and recipient must be identical by the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA-DQB1.
* Peripheral blood stem cells or bone marrow as a graft source
* Diagnosis:

Acute myeloid leukemia Chronic myeloid leukemia, Ph+ Myelodysplastic Syndromes Myeloprolipherative neoplasms - High-risk disease defined as: Acute myeloid leukemia: >5% of clonal blasts in bone marrow despite adequate previous induction therapy or allogeneic stem cell transplantation Myelodysplastic Syndrome: >5% of blasts despite previous therapy Myeloid malignancy with with -7 or complex karyotype, or p53 mutation regardless of blast count in bone marrow Treatment-related myelodysplastic syndrome Second or subsequent allogeneic HCT after relapse of a myeloid malignancy Chronic myelomonocytic leukemia Myeloprolipherative neoplasms, unclassifiable

- No severe concurrent illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2026-12-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival analysis | 2 years
  Measure: Kaplan-Meier estimate of death from all causes

SECONDARY OUTCOMES:
Incidence of secondary hemophagocytic lymphohistiocytosis | 100 days
  Based on H-score diagnostic criteria.
Incidence of HSCT-associated adverse events (safety and toxicity) | 100 days
  Toxicity assessment is based on NCI CTC AE 6.0 grades. Veno-occlusive disease incidence and severity assessment is based on EBMT criteria 2016. Transplant-associated microangiopathy incidence assessment is based on Schoettler et al. criteria. All toxicity measurements will be aggregated as severity scores.
Infectious complications, including analysis of severe bacterial, fungal and viral infections incidence | 100 days
  Proportion of patients, requiring systemic treatment for bacterial, viral and fungal disease
Incidence of acute GVHD grade II-IV | 180 days
  Cumulative incidence of patients with acute GVHD II-IV grade
Incidence of moderate and severe chronic GVHD | 2 years
  Cumulative incidence of patients with moderate and severe chronic GVHD according to MAGIC 2018 criteria
Non-relapse mortality analysis | 2 years
  Cumulative incidence of patients with mortality without hematological relapse of malignancy
Relapse rate analysis | 2 years
  Cumulative incidence of patients with relapse
Event-free survival analysis | 2 years
  Kaplan-Meier estimate of death or relapse
GVHD-event-free survival analysis | 2 years
  Kaplan-Meier estimate of death, grade III-IV acute GVHD, severe chronic GVHD or relapse

CONTACTS AND LOCATIONS:
Locations (1):
- Pavlov University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 10 years
Access Criteria: Submit a study proposal and request to use the data to Pavlov University Clinical Trial department: spbgmutrials@yandex.ru

REFERENCES:
- [Background] Moiseev I, Bondarenko S, Vlasova Y, Morozova E, Smirnova A, Epifanovskaya O, Zhogolev D, Chernishova D, Meliboev A, Khudayberdiev J, Mazing A, Lapin S, Kholopova I, Botina A, Baykov V, Popova M, Kosarev O, Kulagin A. Allogeneic hematopoietic cell transplantation with a combination of posttransplantation bendamustine and cyclophosphamide in refractory myeloid neoplasms. Cancer. 2025 May 15;131(10):e35893. doi: 10.1002/cncr.35893. PMID 40372957